CLINICAL TRIAL: NCT05815771
Title: Clinical and Magnetic Resonance Imaging Evaluation of Micro Fragmented Adipose Tissue Injection Combined With Bone Marrow Stem Cells on Healing of Temporomandibular Joint Internal Disc Derangement Without Reduction (Randomized Control Pilot Clinical Trial)
Brief Title: Clinical and Magnetic Resonance Imaging Evaluation of Micro Fragmented Adipose Tissue Injection Combined With Bone Marrow Stem Cells on Healing of Temporomandibular Joint Internal Disc Derangement Without Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mohamed Talaat Abbas Hassan (Other)
Responsible Party: Sponsor-Investigator, Mohamed Talaat Abbas Hassan, Principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stem cells injection of TMJ
Record Dates: First submitted 2023-03-13; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Micro fragmented adipose tissue (Active Comparator): Micro fragmented adipose tissue mixed with Bone marrow stem cells injection on healing of TMJ internal disc derangement without reduction
  Interventions: Procedure: Micro fragmented adipose tissue mixed with bone marrow stem cells; Procedure: Bone Marrow stem cells aspirate
- Bone marrow stem cells aspiration (Active Comparator): Bone marrow stem cells injection on healing of TMJ internal disc derangement without reduction
  Interventions: Procedure: Micro fragmented adipose tissue mixed with bone marrow stem cells; Procedure: Bone Marrow stem cells aspirate
- hyaluronic acid gel injection (Placebo Comparator): Intra and periarticular injection of 2 mm of hyaluronic acid gel on healing of TMJ internal disc derangement without reduction
  Interventions: Procedure: Micro fragmented adipose tissue mixed with bone marrow stem cells; Procedure: Bone Marrow stem cells aspirate

INTERVENTIONS:
Procedure: Micro fragmented adipose tissue mixed with bone marrow stem cells — mixture of stem cells
Procedure: Bone Marrow stem cells aspirate — stem cells

SUMMARY:
Arthrocentesis of TMJ then injection of micro fragmented adipose tissue mixed with bone marrow aspirate on healing of TMJ internal disc derangement without reduction.

DETAILED DESCRIPTION:
Arthrocentesis of TMJ then injection of intra and periarticular of 2 mm of micro fragmented adipose tissue mixed with Bone marrow aspirate extracted from 20 mm of bone marrow using gradient separation method in one group and use of Bone marrow aspirate injection only in another group and injection of intra and periarticular of 2 mm hyaluronic acid gel in control group on healing of TMJ internal disc derangement without reduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with TMDs not previously surgically treated.
* Patients with TMJ osteoarthritis assessed by clinical examination and magnetic resonance imaging.

Exclusion Criteria:

* Patients refuse to be enrolled in this study.
* Patients with uncontrolled systemic disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Mandibular mouth opening | 6 Months
  Measuring Maximum interincisal opening measured by plastic scale ruler in millimeter

SECONDARY OUTCOMES:
Post-operative pain | six months follow-up
  measuring pain by using visual analogue scale from (0 to 10) score where zero indicate no pain and 10 indicate worst pain
Joint sound | six months follow-up
  Clicking by clinical examination indicate ( present or absent ) of clicking
Lateral and protrusive movements | six months follow-up
  Measuring lateral and protrusive movements by using range of motion scale in millimeter

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo university, Cairo
  - Mohamed Talaat Abbas Hassan, Cairo